CLINICAL TRIAL: NCT02868177
Title: Totum-63 Effect on Glucose and Lipid Homeostasis in People With Abdominal Obesity Associated With Impaired Glucose Tolerance or Untreated Type 2 Diabetes and Hypertriglyceridemia
Brief Title: Effect of Totum-63, Active Ingredient of Valedia, on Glucose and Lipid Homeostasis on Subjects With Prediabetes
Acronym: TOTUM-63 TWO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other); Institut Pasteur de Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-A00484-47
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Prediabetes; Type 2 Diabetes; Hypertriglyceridemia; Obesity; Disease; Insulin Resistance
Keywords: Prevention
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Hypertriglyceridemia; Obesity; Disease; Insulin Resistance | interventions — TOTUM-63

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Totum-63 (Experimental): The studied active product is a food supplement formula in shape of capsule which contains Totum-63 (a patented mixture of dry extracts from 5 plants), active ingredient of Valedia
  Interventions: Dietary Supplement: Totum-63
- Placebo (Placebo Comparator): The comparative product is a placebo with the same characteristics of appearance and packaging in which all ingredients are replaced by maltodextrin.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Totum-63 — Each randomized subject will consume 8 capsules daily of either active (5200 mg of Totum-63) during 24 weeks (from visit V1 to visit V3). They will consume 3 capsules at the beginning of their breakfast, 2 capsules at the beginning of their lunch and 3 capsules at the beginning of their dinner.
  Arms: Totum-63
Dietary Supplement: Placebo — Each randomized subject will consume 8 capsules daily of placebo (5064 mg of maltodextrine) during 24 weeks (from visit V1 to visit V3). They will consume 3 capsules at the beginning of their breakfast, 2 capsules at the beginning of their lunch and 3 capsules at the beginning of their dinner.
  Arms: Placebo

SUMMARY:
Given the data on the active ingredients of Totum-63, this research aims to evaluate the effect of its chronic consumption (24 weeks) on glucose and lipid homeostasis and especially on fasting plasma glucose in volunteers with abdominal obesity associated with impaired glucose tolerance or untreated type 2 diabetes and hypertriglyceridemia. This clinical study is designed to estimate the effect of Totum-63, active ingredient of Valedia, on several glucose and lipid homeostasis related parameters since these data are still unknown for this specific dietary supplement formula. Collected data will provide more reliable information which may be used to plan a subsequent larger main study.

DETAILED DESCRIPTION:
Primary objective:

The primary objective of the present trial is to assess the beneficial effect of Totum-63 compared to a placebo on glucose homeostasis assessed by the fasting plasma glucose level in prediabetics or untreated type 2 diabetics after 24 weeks of consumption.

Secondary objectives:

Secondary objectives of the study are to assess the efficacy of Totum-63 compared to a placebo in prediabetics or untreated type 2 diabetics after 12 and 24 weeks of consumption through the following criteria:

* Glucose homeostasis assessed by fasting plasma glucose level (after 12 weeks of consumption only), fasting blood HbA1c and fructosamine levels, OGTT (Oral Glucose Tolerance Test after 24 weeks of consumption only), insulinemic and glycemic parameters.
* Pancreatic beta-cells function and insulin sensitivity assessed by fasting blood insulin level, HOMA-IR (Homeostasis Model Assessment of Insulin Resistance), HOMA-β, QUICKI (Quantitative Insulin sensitivity Check Index), ISI-M (Matsuda-DeFronzo Insulin Sensitivity Index after 24 weeks of consumption only), OGIS (Oral Glucose Insulin Sensitivity after 24 weeks of consumption only) and PREDIM (PREDIcted M after 24 weeks of consumption only) indexes.
* Lipid homeostasis assessed by fasting blood levels of triglycerides (TG), Total Cholesterol (TC), HDL-cholesterol, LDL-cholesterol and NEFA (Non-Esterified Fatty Acids).
* Oxidation mechanism of circulating lipids assessed by the ratio fasting blood LDLox / fasting blood LDLc and the PON-1 (paraoxonase-1, arylesterase activity) activity in blood.
* Low grade inflammation assessed by fasting blood hsCRP level.
* Hepatic function assessed by fasting blood total bilirubin level, GGT, ASAT and ALAT activities in blood.
* Hemodynamics assessed by Heart Rate (HR), Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP).
* Anthropometrics assessed by Body Weight (BW), Waist Circumference (WC), Hip Circumference (HC) and Waist to Hip Ratio (WHR).
* Satiety assessed by the three-day food diary energy and nutrient intake parameters.

Safety objectives:

The following criteria assessed after 24 weeks of study product consumption participate to the objectives of safety check:

* Renal function assessed by fasting blood creatinine and urea level;
* Complete blood count.

ELIGIBILITY:
Inclusion Criteria:

I1. Fasting glycemia > 6,1 mmol/L. (1,1 g/L). I2. 2 hours glycemia (OGTT) > 7,8 mmol/L (1,4 g/L). I3. HbA1c < 7% I4. Triglyceridemia > 1,5 g/L. I5. Prediabetic or type-2 diabetic but not requiring immediate drug therapy according to the current recommendations (HAS, 2013).

I6. Waist circumference > 94 cm for men or > 80 cm for women. I7. With reported body weight variation < 5% in the 3 months prior the randomization.

I8. Without significant change in food habits or in physical activity in the 3 months before randomization and agreeing to keep them unchanged throughout the study (no hyper-hypocaloric diet nor start-stop of sport activity planned in the next 7 months).

I9. For women: Non menopausal with the same reliable contraception since at least three months before the beginning of the study and agreeing to keep it during the entire duration of the study (hormonal contraception, intra uterine device or surgical intervention) or menopausal with or without hormone replacement therapy (oestrogenic replacement therapy begun from less than 3 months excluded).

I10. Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination.

I11. Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form.

I12. Affiliated with a social security scheme. I13. Agree to be registered on the volunteers in biomedical research file.

Exclusion Criteria:

E1. Fasting blood triglycerides > 3,5 g/L. E2. TSH outside the laboratory normal values. E3. Fasting blood TC > 4,5 g/L or HDLc < 0,1 g/L with an abnormality judged as clinically significant according to the investigator.

E4. Blood AST, ALT or GGT > 3xULN (laboratory Upper Limit of Normal). E5. Blood urea > 12 mmol/L or creatinine > 125 µmol/L. E6. Complete blood count with hemoglobin < 11 g/L or leucocytes < 3000 / mm3 or leucocytes > 16000 / mm3 or clinically significant abnormality according to the investigator.

E7. Suffering from a metabolic disorder such as treated diabetes, uncontrolled thyroidal trouble or other metabolic disorder.

E8. Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg).

E9. With a history of retinopathy, microalbuminuria, ischemic cardiovascular event or, during the previous 6 months a surgical procedure.

E10. Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease).

E11. Under antidiabetic drug (e.g. biguanides, sulfonylureas, glinides, gliptines, glitazones, gliflozines, α-glucosidase inhibitors, incretins and insulin).

E12. Under lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 3 months before the randomization.

E13. Requiring cholesterol lowering by immediate pharmacologic intervention according to the current recommendations (AFSSAPS 2005).

E14. Under medication which could affect glucose and/or lipid homeostasis parameters or stopped less than 3 months before randomization (e.g. beta 2 agoniste like salbutamol, Angiotensin Converting Enzyme (ACE) inhibitors, beta blockers, thiazide diuretics, Selective Serotonin Reuptake Inhibitors (SSRIs), Mono-Amine Oxidase Inhibitors (MAOIs), neuroleptics, long-term corticosteroid systemic drugs, systemic antibodies, androgens, phenytoin, interferons, immunosuppressants, antivirals and antiretrovirals, etc.). Beta 2 agoniste like salbutamol, ACE inhibitors, beta blockers, thiazide diuretics, SSIRs, MAOIs begun more than 3 months before the randomization and maintained stable during the whole study are tolerated. The others drugs (neuroleptics, long-term corticosteroid systemic drugs, systemic antibodies, androgens, phenytoin, interferons, immunosuppressants, antivirals and antiretrovirals, etc.) are not allowed during the study.

E15. Regular intake of dietary supplements or "health foods" rich in plant stanol or sterol (like PRO-ACTIV or DANACOL products), in long chain omega-3 fatty acids (especially sofgels containing fish oils), or in other substances intended to lower LDLc, TG or glycemia (e.g. beta-glucans, konjac, cinnamon, olive leaf extract, berberine, red yeast rice, policosanol, etc.) or stopped less than 3 months before the randomization.

E16. Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the randomization.

E17. Under dietary supplement in the month before V1. E18. With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient.

E19. Consuming more than 3 standard drinks of alcoholic beverage for men or 2 standard drinks daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study.

E20. With extreme eating habits (e.g. vegetarian or vegan). E21. With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator.

E22. Smoking more than 10 cigarettes daily or not agreeing to keep his smoking habits unchanged throughout the study.

E23. Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded).

E24. Pregnant or lactating women or intending to become pregnant within 7 months ahead.

E25. Who made a blood donation in the 3 months before the randomization or intending to make it within 7 months ahead.

E26. Taking part in another clinical trial or being in the exclusion period of a previous clinical trial.

E27. Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros.

E28. Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision.

E29. Presenting a psychological or linguistic incapability to sign the informed consent.

E30. Impossible to contact in case of emergency.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Changes in fasting glycemia | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in g/L

SECONDARY OUTCOMES:
Changes in fasting glycemia | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood levels of HbA1c | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in %
Changes in fasting blood levels of HbA1c | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in %
Changes in fasting blood levels of fructosamine | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in µmol/L
Changes in fasting blood levels of fructosamine | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µmol/L
Changes in fasting insulinemia | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in mU/L
Changes in fasting insulinemia | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mU/L
Changes in the evolution of glycemia during an oral glucose tolerance test | 24 weeks
  Changes between V1 (baseline) and V3 (24 weeks) visits (defined as the difference V3-V1 in g/L) of glycemia at 30, 60, 90 and 120 minutes, glucose Cmax and Δpeak (difference from the baseline at Cmax) and Incremental Area Under the Curve (iAUC) of glycemia between T0 and T120 minutes following the 75g glucose intake (iAUC0-120min) and considering the following time-points: T0, T30, T60, T90 and T120
Changes in the evolution of insulinemia during an oral glucose tolerance test | 24 weeks
  Changes between V1 (baseline) and V3 (24 weeks) visits (defined as the difference V3-V1 in g/L) of insulinemia at 30, 60, 90 and 120 minutes, insulin Cmax and Δpeak (difference from the baseline at Cmax) and Incremental Area Under the Curve (iAUC) of insulinemia between T0 and T120 minutes following the 75 g glucose intake (iAUC0-120min) and considering the following time-points: T0, T30, T60, T90 and T120
Changes in HOMA-IR, HOMA-β, QUICKI, ISI-M, OGIS and PREDIM indices | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline)
Changes in HOMA-IR, HOMA-β and QUICKI indices | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline)
Changes in fasting blood concentrations of triglycerides, non esterified fatty acids, LDL cholesterol, HDL cholesterol and Total cholesterol | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of triglycerides, non esterified fatty acids, LDL cholesterol, HDL cholesterol and Total cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood level of PON-1 (Paraoxonase) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in μkat/L
Changes in fasting blood level of PON-1 (Paraoxonase) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in μkat/L
Changes in the ratio of fasting blood oxidized LDL / fasting blood LDL cholesterol | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in U/g
Changes in the ratio of fasting blood oxidized LDL / fasting blood LDL cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in U/g
Changes in fasting blood level of hsCRP | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in mg/L
Changes in fasting blood level of hsCRP | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mg/L
Changes in fasting blood levels of ASAT (Aspartate aminotransferase) and ALAT (Alanine aminotransferase) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood levels of GGT (Gamma glutamyltransferase) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood levels of bilirubin | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in µmol/L
Changes in fasting blood levels of creatinine | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in µmol/L
Changes in fasting blood levels of creatinine | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µmol/L
Changes in heart rate | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in bpm
Changes in heart rate | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in bpm
Changes in SBP (systolic blood pressure) and DBP (diastolic blood pressure) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in mmHg (mean of the two measures for each parameter at each visit)
Changes in SBP (systolic blood pressure) and DBP (diastolic blood pressure) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mmHg (mean of the two measures for each parameter at each visit)
Changes in body weight | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in kg
Changes in body weight | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in kg
Changes in WC (waist circumference) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in cm
Changes in WC (waist circumference) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in cm
Changes in HC (hip circumference) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in cm
Changes in HP (hip circumference) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in cm
Changes in WHR (waist to hip ratio) | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline)
Changes in WHR (waist to hip ratio) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline)

OTHER OUTCOMES:
Changes in total energy intake | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in kcal/day (mean of the 3 days of the food diary)
Changes in total energy intake | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in kcal/day (mean of the 3 days of the food diary)
Changes in percentage of energy intake from fat, carbohydrates and protein | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in % (mean of the 3 days of the food diary)
Changes in percentage of energy intake from fat, carbohydrates and protein | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in % (mean of the 3 days of the food diary)
Changes in saturated fatty acids intake | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in g (mean of the 3 days of the food diary)
Changes in saturated fatty acids intake | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g (mean of the 3 days of the food diary)
Changes in physical activity score | 24 weeks
  Defined as the difference V3 (24 weeks) - V1 (baseline) in MET-min/week (assessed by IPAQ SF)
Changes in physical activity score | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in MET-min/week (assessed by IPAQ SF)

CONTACTS AND LOCATIONS:
Overall Officials: David GENDRE, Dr, Principal Investigator — Biofortis Mérieux NutriSciences; Sébastien L PELTIER, PhD, Study Director — Valbiotis; Jean-Marie BARD, Dr-PhD, Study Chair — UFR des Sciences Pharmaceutiques et Biologiques, Nantes, France
Locations (6):
- France (2):
  - Institut Pasteur de Lille, Lille
  - Biofortis Mérieux NutriSciences Clinical Investigation Center, Saint-Herblain
- Atlantia Food Clinical Trials, Cork, Ireland
- Serbia (2):
  - Clinical center of Kragujevac, / Poseidon CRO, Kragujevac
  - Clinical Center of Vojvodina / Poseidon CRO, Novi Sad
- University Medical Centre Ljubljana / Poseidon CRO, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided